CLINICAL TRIAL: NCT03222739
Title: Slicer+PLUS: Collaborative, Open-source Software for Ultrasound Analysis
Brief Title: Ultrasound for Scoliosis Diagnostic Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's National Research Institute (Other)
Collaborators: Kitware, Inc. (Unknown); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Kevin Cleary, Technical Director, Bioengineering Initiative, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro8456; R01EB021396-01A1 (NIH)
Record Dates: First submitted 2017-07-13; First posted 2017-07-19 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Juvenile
MeSH Terms: conditions — Scoliosis | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: A single-arm unblinded group of patients will receive ultrasound imaging of spine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device Arm (Other): This is a single arm study comparing an ultrasound with the industry standard of x-ray to detect and monitor scoliosis curvature.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — An industry standard ultrasound will be fitted with a self-tracking probe to track along the spine. The ultrasound will be performed three (3) times along the spine at initial consultation for scoliosis.

SUMMARY:
Scoliosis is a complex 3-dimensional deformity of the spine. It may occur at any time throughout growth and development and is typically detected through x-ray imaging. Although effective at visualizing a curve, x-ray imaging is costly and may expose children to potentially harmful ionizing radiation. This is a 30 patient study to evaluate the reliability of ultrasound, an imaging technique without radiation, to effectively measure scoliosis deformities compared to the gold-standard of x-ray.

DETAILED DESCRIPTION:
All patients who present to Children's National Medical Center for initial evaluation of idiopathic or juvenile scoliosis will be approached.

ELIGIBILITY:
Inclusion Criteria:

* All patients ages 7-17 years who present to Dr. Matthew Oetgen in the Department of Orthopaedic Surgery & Sports Medicine for clinical evaluation of scoliosis,
* Scoliosis curve type to include adolescent idiopathic (AIS) or juvenile, and
* Have x-rays taken as part of clinical evaluation

Exclusion Criteria:

* Not willing or able to provide consent, or
* Had x-rays taken at an outside facility, or
* Any underlying neuromuscular condition or syndrome and congenital deformities

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-03-14 (Actual); Primary Completion 2023-12-06 (Estimated); Study Completion 2023-12-06 (Estimated)

PRIMARY OUTCOMES:
Imaging | 3 years
  Ability of the ultrasound to produce a radiographic measurement (e.g. coronal spinal curvature, coronal spinal rotation) within the variability of the gold standard of x-ray

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States